CLINICAL TRIAL: NCT01224613
Title: A Randomized Controlled Trial To Compare The Immunogenicity Of Self-Administered And Nurse-Administered Intradermal Influenza Vaccine
Brief Title: Study to Compare Self-administered and Nurse-administered Intradermal Influenza Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: IWK Health Centre (Other); MCM Vaccines B.V. (Industry); Mount Sinai Hospital, Canada (Other)
Responsible Party: Shelly McNeil, Canadian Center for Vaccinology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SP1002
Record Dates: First submitted 2010-10-14; First posted 2010-10-20 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intanza - self-administered (Active Comparator): Self-administered intradermal influenza vaccine
  Interventions: Biological: Intanza
- Intanza - nurse-administered (Active Comparator): Nurse-administered intradermal influenza vaccine
  Interventions: Biological: Intanza

INTERVENTIONS:
Biological: Intanza — 0.1 mL of Intanza intradermally at visit # 1
  Other Names: Influenza Vaccine (Split Virion, Inactivated)
  Arms: Intanza - self-administered
Biological: Intanza — 0.1 mL of Intanza intradermally at visit #1
  Other Names: Influenza Vaccine (Split Virion, Inactivated)
  Arms: Intanza - nurse-administered

SUMMARY:
The purpose of this study is to compare the immunogenicity and reactogenicity of self-administered intradermal influenza vaccine (Intanza)to nurse-administered.

DETAILED DESCRIPTION:
Participants will be randomized at visit one to either receive self-administered or nurse-administered intradermal influenza vaccine (Intanza). A blood sample will be taken prior to vaccination and 21 days post-vaccination. Participants will record information in a memory aid for 7 days including daily temperatures, solicited, unsolicited and general reactions. They will be called on study Day 8 to collect this information. Participants will return 21-24 days later for follow-up serology and review of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable persons between age of 18-60
* Available during the trial period and for follow-up
* Able to read, understand, and sign informed consent
* Able to be contacted by telephone for follow-up of adverse events

Exclusion Criteria:

* Use of experimental vaccines within the month prior to study entry, or expected use of experimental or licensed vaccines or blood/blood products during the duration of the study.
* Receipt of immunoglobulin or other blood product within 3 months prior to enrollment
* Receipt of other licensed vaccines within the preceding 4 weeks
* History of a severe reaction following influenza vaccination
* Use of cytotoxic therapy or biologic modifiers in the previous 2 years.
* Plans to receive cytotoxic therapy during the study period.
* Concurrent acute moderate to severe illness. (Vaccination will be deferred until recovery. Subjects with mild illnesses with fever ≤37.8ºC orally may be enrolled).
* History of medical disorder associated with immunosuppression (eg. including HIV-infected individuals, transplant recipients)
* History of chronic lung, cardiac, renal or liver disease, which has required hospitalization in the last year.
* Receipt of any high-dose daily systemic corticosteroids (inhaled steroids are acceptable) within two weeks of study entry. High dose is defined as a dose of 20 mg of prednisone daily or its equivalent. Topical steroids are allowed.
* Failure to give written, informed consent
* History of febrile illness (>37.8ºC orally) within the past 72 hours (immunization may be deferred).
* Known allergy to eggs or other components of vaccine (i.e., thimerosal)
* History of Guillain-Barré Syndrome (GBS)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 276 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | 21 days post-vaccination
  That the immunogenicity of self-administered intradermal 2010/11 seasonal influenza vaccine (Intanza) is non-inferior to that of nurse administered intradermal 2010/11 seasonal influenza vaccine. Specifically, that ratio of increase in geometric mean titres between day 0 and day 21 post-vaccination are greater than 2/3 (i.e. GMT (IDS)/GMT (IDN) > 0.65).

SECONDARY OUTCOMES:
Reactogenicity | 7 days post-vaccination
  The reactogenicity of self-administered intradermal 2010/11 seasonal influenza vaccine (Intanza) is not significantly greater than that of nurse administered intradermal 2010/11 seasonal influenza vaccine.
Observational | at vaccination
  85% or more of healthy adults can self-administer Intanza successfully; that is, they are willing to self-administer vaccine and successfully administer it, as judged by observation by a trained nurse.

CONTACTS AND LOCATIONS:
Overall Officials: Shelly McNeil, MD, Principal Investigator — Canadian Center for Vaccinology
Locations (2):
- Canada (2):
  - Canadian Center for Vaccinology, Halifax, Nova Scotia
  - Mount Sinai Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Coleman BL, McGeer AJ, Halperin SA, Langley JM, Shamout Y, Taddio A, Shah V, McNeil SA. A randomized control trial comparing immunogenicity, safety, and preference for self- versus nurse-administered intradermal influenza vaccine. Vaccine. 2012 Sep 28;30(44):6287-93. doi: 10.1016/j.vaccine.2012.08.006. Epub 2012 Aug 16. PMID 22902784